CLINICAL TRIAL: NCT04752384
Title: Transdermal Buprenorphine for the Treatment of Radiation-Induced Mucositis Pain in Head and Neck Cancer Patients: A Pilot Study
Brief Title: Transdermal Buprenorphine for the Treatment of Radiation-Induced Mucositis Pain in Head and Neck Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Stuart Wong, Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PRO00040100
Record Dates: First submitted 2021-02-10; First posted 2021-02-12 (Actual); Results first posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: Mucositis; Radiation; Chemoradiation; visual analog scale; Buprenorphine; Tramadol; Brief Pain Inventory; Oral Mucositis Pain App
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Mucositis | interventions — Buprenorphine; Tramadol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Drug Treatment (Experimental): The main objective of this study is to provide preliminary evidence that FDA approved dose of transdermal buprenorphine in conjunction with oral tramadol can provide adequate analgesia of radiation-induced mucositis pain during treatment and follow up period in head and neck cancer patients.
  Interventions: Drug: Buprenorphine; Drug: Tramadol; Device: Oral Mucositis (OM) Pain App

INTERVENTIONS:
Drug: Buprenorphine — Transdermal buprenorphine will be started at 5 mcg/hr once a week. Depending on the Visual Analog Scale (VAS) score, it may be increased up to 20 mcg/hr once a week.
  Other Names: Belbuca; Probuphine; Buprenex
Drug: Tramadol — Oral tramadol will be started at 50 mg/day. Depending on the Visual Analog Scale (VAS) score, it may be increased up to 400 mg/day.
  Other Names: Ultram; Ryzolt; ConZip
Device: Oral Mucositis (OM) Pain App — Each study participant will be issued an Android smartphone, or he or she may use his/her own compatible device (whether or not it has an active data service) to which the OM Pain App will be downloaded and installed. Subjects will receive a preprogrammed alarm four times a day from their smartphones prompting them to directly enter OM pain levels on the device. Patients may submit as many pain entries as they wish beyond the four minimum levels.
  Subjects will receive a preprogrammed alarm four times a day from their smartphones prompting them to directly enter OM pain levels on the device. Patients may submit as many pain entries as they wish beyond the four minimum levels.
  Other Names: OM Pain App

SUMMARY:
This is a single-arm prospective clinical trial to determine the safety and feasibility of using transdermal buprenorphine in alleviation of radiation induced mucositis pain in head and neck cancer patients.

DETAILED DESCRIPTION:
Hypothesis: Long-acting transdermal buprenorphine (FDA-approved dose from 5 mcg to 20 mcg /week) in conjunction with oral tramadol (50mg-400mg) as needed for breakthrough pain would lead to significant reduction in mucositis-related pain in locally advanced head and neck cancer patients being treated with radiation therapy by the end of treatment and follow up period of 12 weeks.

This is a single-arm, interventional, supportive care clinical trial for head and neck cancer patients evaluating role of transdermal (TD) buprenorphine and tramadol combination in alleviating radiation-induced mucositis pain. This will generate preliminary data to test the feasibility and efficacy of study drug regimen. The study will also test the clinical usefulness of the smart phone pain app in recording and reporting radiation induced mucositis pain.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-80 years.
2. Histologically confirmed malignancies involving the oral cavity, oropharynx, hypopharynx and larynx (including non-squamous cell histologies, salivary gland carcinomas and unknown primary tumors).
3. Undergoing a course of either definitive radiation (dose of at least 50 Gy to the head and neck region) +/-chemotherapy or adjuvant radiation (at least 50 Gy to the head and neck region) +/- chemotherapy (Patients with a history of prior definitive course of radiation will be allowed).
4. Eastern Cooperative Oncology Group (ECOG) Performance status ≤ 2
5. Concurrent enrollment on interventional trial is allowed.
6. English speaking and literate
7. Patients will be allowed to take radiotherapy mix, viscous lidocaine or magic mouthwash like agents that do not contain opioids. Tylenol allowed for fever and mild pain before starting drug regimen.
8. Adequate organ function: Minor dose adjustments for tramadol is required in severe liver and renal impairment so we would only include patients with adequate organ function outlined in below. No dose adjustment for renal or hepatic impairment is required for TD buprenorphine. Some other parameters like hemoglobin, platelets and white blood count (WBC) are required for administration of standard of care chemotherapy like cisplatin along with radiation in treatment of head and neck squamous cell carcinoma (HNSCC). They are not required for administration of buprenorphine or tramadol.

   1. total bilirubin < 2 mg/dL
   2. aspartate aminotransferase (AST) / alanine aminotransferase (ALT) < 5 times institutional upper limit
   3. creatinine clearance > 30 mL/min/1.73 m2 for patients with creatinine levels above institutional normal"
9. Pregnancy: It is known that standard of care treatments of HNSCC radiation therapy and chemotherapy have detrimental effects on human pregnancy or development of the embryo or fetus. Therefore, female patients participating in this study should avoid becoming pregnant, and male patients should avoid impregnating a female partner. Non-sterilized female patients of reproductive age and male patients should use effective methods of contraception through defined periods during and after study treatment as specified below.

   Female patients must meet one of the following:
   * Postmenopausal for at least one year before the screening visit, or
   * Surgically sterile, or
   * If they are of childbearing potential, agree to practice two effective methods of contraception from the time of signing of the informed consent form through three months after the last dose of study drug, AND
   * Must also adhere to the guidelines of any treatment-specific pregnancy prevention program, if applicable, or
   * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post ovulation methods] and withdrawal are not acceptable contraception methods.)

   Male patients, even if surgically sterilized (i.e., status post vasectomy), must agree to one of the following:
   * Practice effective barrier contraception during the entire study treatment period and through 90 days after the last study drug dose, OR
   * Must also adhere to the guidelines of any treatment-specific pregnancy prevention program, if applicable, OR
   * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post ovulation methods] and withdrawal are not acceptable methods of contraception.)
10. Ability to understand a written informed consent document, and the willingness to sign it.
11. Possession of a smart phone (android or apple-based platforms) and ability to operate a smart phone application. Patients who do not have smart phones will be provide wireless devices that have OM pain app installed on them.

Exclusion Criteria:

1. Physical exam demonstrating preexisting mucositis.
2. Preexisting oral infection or ongoing toxicity from prior radiotherapy.
3. History of substance abuse, positive urine drug screen in last six months.
4. Patients with multiple distant metastasis (subjects with resectable oligometastasis will be allowed)
5. Current or recent use (within four weeks of screening) of mixed opioid agonists/antagonists or other opioid antagonists. Methadone use within four weeks of screening.
6. History of prolonged QTc>greater than 450 milliseconds in males and greater than 470 milliseconds in females.
7. Patients on systemic therapy (chemotherapy or immunotherapy) for another cancer subtype.
8. Patients receiving induction chemotherapy prior to or after radiation/chemoradiation like patients with nasopharyngeal carcinoma
9. Patients with history of abdominal surgery within 60 days of registration, acute gastrointestinal conditions like colitis and appendicitis within four weeks of screening.
10. Patients with conditions that may compromise blood-brain barrier permeability. The blood-brain barrier may become leaky in select neurological diseases, such as amyotrophic lateral sclerosis, epilepsy, brain trauma and edema
11. Patients with a history of myocardial infarction ≤ 6 months prior to registration.
12. Patients with h/o significant respiratory depression; acute or severe bronchial asthma; known or suspected gastrointestinal obstruction, including paralytic ileus.
13. History of serious or severe hypersensitivity reaction to buprenorphine or tramadol or any of its excipients.
14. Patients on anti-depressant and anti-psychotic therapy
15. Pregnant and lactating women are excluded from this study because chemotherapy and radiation given for treatment of HNSCC has a potential for teratogenic or abortifacient effects. Additionally, Buprenorphine is classified as category C for use during pregnancy, which means that the risk of adverse effects on the fetus cannot be ruled out. Buprenorphine does cross the placenta, and the use of opioids during pregnancy may result in neonatal withdrawals soon after birth. Symptoms of this may include irritability, apnea, increased tone, tremor, convulsions, or respiratory depression in the neonate. The onset of withdrawal in a neonate whose mother has taken buprenorphine during the pregnancy could be anywhere from the first day of life to the eighth day of life.
16. Patients with history of seizure disorder as oral tramadol may reduce seizure threshold.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-07-08 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2024-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart J. Wong, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert & the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Drug Treatment: The main objective of this study is to provide preliminary evidence that FDA approved dose of transdermal buprenorphine in conjunction with oral tramadol can provide adequate analgesia of radiation-induced mucositis pain during treatment and follow up period in head and neck cancer patients.
  Buprenorphine: Transdermal buprenorphine will be started at 5 mcg/hr once a week. Depending on the Visual Analog Scale (VAS) score, it may be increased up to 20 mcg/hr once a week.
  Tramadol: Oral tramadol will be started at 50 mg/day. Depending on the Visual Analog Scale (VAS) score, it may be increased up to 400 mg/day.
  Oral Mucositis (OM) Pain App: Each study participant will be issued an Android smartphone, or he or she may use his/her own compatible device (whether or not it has an active data service) to which the OM Pain App will be downloaded and installed. Subjects will receive a preprogrammed alarm four times a day from their smartphones prompting them to directly enter OM pain levels on the device. Patients may submit as many pain entries as they wish beyond the four minimum levels.
  Subjects will receive a preprogrammed alarm four times a day from their smartphones prompting them to directly enter OM pain levels on the device. Patients may submit as many pain entries as they wish beyond the four minimum levels.
Period: Overall Study
Arm/Group | Drug Treatment
Started | 20
Completed | 18
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Drug Treatment
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: The Number of Subjects Who Achieve at Least a 30 Percent Decrease in Pain From Baseline in VAS Pain Score Calculated From BPI Questionnaire.
Description: The Brief Pain Inventory - Short Form (BPI-sf) is a nine-item self-administered questionnaire used to evaluate the severity of a patient's pain and the impact of this pain on the patient's daily functioning. The patient is asked to rate their worst, least, average, and current pain intensity -- 0 being no pain and 10 being the pain as bad as you can imagine (within the previous 24 hours).
Time Frame: Baseline up to Week 9
Population: Please note there were many subjects who did not fill out forms.
Measure: Count of Participants; unit: Participants
Arm/Group | Drug Treatment
Number analyzed (Participants) | 13
Participants | 8

2. Secondary Outcome: The Number of Subjects Who Achieve at Least a 30 Percent Decrease in Pain From Baseline in Average Daily Pain Score Calculated by OM Pain App.
Description: The Oral Mucositis (OM) Pain App is a smartphone application that was designed to permit subjects to key in pain severity using a visual analog 0-10 scale. The amount of pain that a subject feels ranges across a continuum from none (0) to an extreme amount of pain (10). The App is programed with an alarm to prompt the patient to record pain severity at prescribed intervals daily and through spontaneous patient input. Compliance is measured by subjects entering in a value four times a day into the OM Pain App.
Time Frame: Baseline up to Week 9
Population: Many subjects did not wear the OM Pain App.
Measure: Count of Participants; unit: Participants
Arm/Group | Drug Treatment
Number analyzed (Participants) | 9
Participants | 3

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: regular investigator assessment, regular laboratory testing
Arm/Group | Drug Treatment
All-Cause Mortality (participants affected / at risk) | 5/20
Serious Adverse Events (participants affected / at risk) | 4/20
Other Adverse Events (participants affected / at risk) | 19/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug Treatment (N=20)
oral pain (Gastrointestinal disorders) | 1 (1)
dysphagia (Gastrointestinal disorders) | 2 (3)
anorexia (Metabolism and nutrition disorders) | 3 (4)
weight loss (Investigations) | 2 (3)
hypotension (Vascular disorders) | 1 (1)
dehydration (Metabolism and nutrition disorders) | 1 (1)
hypernatremia (Metabolism and nutrition disorders) | 1 (1)
hypokalemia (Metabolism and nutrition disorders) | 1 (1)
delirium (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug Treatment (N=20)
abdominal pain (Gastrointestinal disorders) | 2 (3)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 6 (8)
Anorexia (Metabolism and nutrition disorders) | 8 (10)
Aphonia (Nervous system disorders) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (3)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (2)
Blood lactate dehydrogenase increased (Investigations) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Chills (General disorders) | 3 (4)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Confusion (Psychiatric disorders) | 2 (4)
Constipation (Gastrointestinal disorders) | 12 (15)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
CPK increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 3 (4)
Dehydration (Metabolism and nutrition disorders) | 8 (9)
Delirium (Psychiatric disorders) | 2 (4)
Depression (Psychiatric disorders) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 11 (13)
Diarrhea (Gastrointestinal disorders) | 6 (6)
Dizziness (Nervous system disorders) | 5 (8)
Dry mouth (Gastrointestinal disorders) | 10 (10)
Dysarthria (Nervous system disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 14 (16)
Dysphagia (Gastrointestinal disorders) | 9 (12)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Ear pain (General disorders) | 2 (2)
Edema limbs (General disorders) | 2 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Facial pain (General disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (4)
Fatigue (General disorders) | 13 (21)
Fecal incontinence (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Thick secretions (Gastrointestinal disorders) | 2 (2)
drooling (Gastrointestinal disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (2)
Hearing impaired (Ear and labyrinth disorders) | 2 (3)
cirrhosis (Hepatobiliary disorders) | 1 (1)
Herpes simplex reactivation (Infections and infestations) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2)
Hypernatremia (Metabolism and nutrition disorders) | 1 (3)
Hypertension (Vascular disorders) | 5 (6)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (8)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (6)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 4 (7)
Hyponatremia (Metabolism and nutrition disorders) | 5 (7)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (2)
Hypotension (Vascular disorders) | 3 (4)
fever blister (Infections and infestations) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lip infection (Infections and infestations) | 1 (1)
Lymphedema (Vascular disorders) | 4 (4)
Lymphocyte count decreased (Investigations) | 5 (10)
Malaise (General disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 13 (20)
thigh pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 13 (17)
Neck edema (General disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Neutrophil count decreased (Investigations) | 3 (6)
Oral dysesthesia (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 7 (12)
Paresthesia (Nervous system disorders) | 5 (6)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Platelet count decreased (Investigations) | 6 (6)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Renal calculi (Renal and urinary disorders) | 1 (1)
Sinus infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Phlegm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Scalp pain (Skin and subcutaneous tissue disorders) | 1 (1)
Head laceration/cuts (Skin and subcutaneous tissue disorders) | 1 (1)
Soft tissue Coccyx injury (Skin and subcutaneous tissue disorders) | 1 (1)
knee abrasion (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 12 (13)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Thrush (Infections and infestations) | 7 (8)
Tinnitus (Ear and labyrinth disorders) | 7 (7)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 7 (10)
Weight loss (Investigations) | 11 (18)
White blood cell decreased (Investigations) | 2 (2)
Wound infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-26): https://cdn.clinicaltrials.gov/large-docs/84/NCT04752384/Prot_SAP_000.pdf
  • Informed Consent Form (2024-01-31): https://cdn.clinicaltrials.gov/large-docs/84/NCT04752384/ICF_001.pdf